CLINICAL TRIAL: NCT07047157
Title: The Effect of Video-Based Virtual Reality Education on Self-Confidence and Motivation in Nursing Students: The Case of Peripheral Venous Catheterization
Brief Title: The Effect of Video-Based Virtual Reality Education on Self-Confidence and Motivation in Nursing Students
Acronym: Video-Based Vi
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Esra Aydın (Other)
Collaborators: Erzincan Binali Yildirim Universitesi (Other); Yuzuncu Yil University (Other)
Responsible Party: Sponsor-Investigator, Esra Aydın, Principal Investigator, Assistant Professor of Nursing, Ataturk University
Organization: Ataturk University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EA-2025-VR01
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Peripheral Venous Catheterization; Nursing Students; Clinical Skills Training; Self-confidence in Clinical Decision Making and Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group - Traditional Education with Demonstration (Active Comparator): Participants in this group will receive traditional face-to-face education accompanied by live demonstration of peripheral venous catheterization (PVC) procedure. The educational content will be the same as the intervention group but delivered without the use of virtual reality (VR) technology.
  Interventions: Behavioral: Traditional Education with Demonstration
- Experimental Group -Video-Based Virtual Reality Education (Experimental): Participants in the experimental group will receive video-based virtual reality (VR) education using a headset. The training provides visual and stepwise instruction on peripheral venous catheterization (PVC).
  Interventions: Behavioral: Video-Based Virtual Reality Education

INTERVENTIONS:
Behavioral: Video-Based Virtual Reality Education — Participants receive VR-based video training using a headset. The content includes step-by-step instruction on peripheral venous catheterization.
  Arms: Experimental Group -Video-Based Virtual Reality Education
Behavioral: Traditional Education with Demonstration — Participants receive traditional face-to-face instruction and live demonstration of peripheral venous catheterization (PVC).
  Arms: Control Group - Traditional Education with Demonstration

SUMMARY:
This study is a randomized controlled, parallel patterned, single-blind experimental study conducted to investigate the effects of video-based virtual reality (VR) training on self-confidence and motivation levels of nursing students regarding peripheral venous catheterization (PVC) skills. The intervention group will receive video-based training via VR headsets, while the control group will be presented with the same content via traditional face-to-face narration and demonstration. Self-confidence and motivation levels before and after the training will be assessed with valid scales. The study is expected to contribute to the development of innovative technology-supported teaching strategies in nursing education.

DETAILED DESCRIPTION:
Note: The current affiliation of the Principal Investigator (Esra Aydın) is Gumushane University. However, due to system limitations, the affiliation may still appear as "Ataturk University".

ELIGIBILITY:
Inclusion Criteria:

* Receiving nursing education at the relevant university
* Agreeing to participate in the study voluntarily

Exclusion Criteria:

* Having received training on peripheral venous catheterization before

Max Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-08 (Estimated)

PRIMARY OUTCOMES:
Self-confidence in peripheral intravenous catheterization | Pre-intervention (Day 1) and post-intervention (Day 2)
  The Peripheral Intravenous Catheterization Self-Confidence Scale will be used to assess nursing students' self-confidence in performing peripheral IV catheter insertion. The scale consists of 15 items, each rated on a 5-point Likert scale. The total score ranges from 15 to 75, with higher scores indicating greater self-confidence.

SECONDARY OUTCOMES:
Change in motivation score regarding peripheral intravenous catheterization | Pre-intervention (Day 1) and post-intervention (Day 2)
  The Instructional Materials Motivation Scale (IMMS) will be used to evaluate nursing students' motivation toward the peripheral intravenous catheterization training material. The scale consists of 33 items, each rated on a 5-point Likert scale. The total score ranges from 33 to 165, with higher scores indicating greater motivation.

CONTACTS AND LOCATIONS:
Locations (1):
- Van Yüzüncü Yıl University, Dursun Odabaş Medical Center, Van, Turkey (Türkiye)